CLINICAL TRIAL: NCT06631079
Title: An Open-label, Phase I/II Multicenter Clinical Trial of NECVAX-NEO1 in Addition to Anti-PD-1 or Anti-PD-L1 Monoclonal Antibody Therapy in Patients With Solid Tumors
Brief Title: Personalised Neoantigen-targeting Cancer Vaccine NECVAX-NEO1 in Anti-PD-1/PD-L1 Therapy in Patients With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NEC Bio B.V (Industry)
Collaborators: NEC Bio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NECVAX-NEO1-02-INT
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NECVAX-NEO1 (Experimental): Oral DNA Vaccine
  Interventions: Biological: NECVAX-NEO1

INTERVENTIONS:
Biological: NECVAX-NEO1 — Bacteria-based orally administered personalised neoantigen-targeting cancer vaccine
  Other Names: Personalised neoantigen-targeting oral DNA cancer vaccine

SUMMARY:
Phase I/II multicenter, open-label, single-arm trial in patients to evaluate the safety and effect of NECVAX-NEO1 administered in combination with PD-1/PD-L1 mABs in patients with solid tumors. Patients with solid tumors who will be treated with approved standard of care (SoC) PD-1 or PD-L1 monoclonal antibody inhibitor therapy, and who after starting treatment with PD-1/PD-L1 inhibitor reached either Stable Disease (SD) or Partial Response (PR) (Cohort 1) or PD (Cohort 2) according to RECIST 1.1 and iRECIST assessed at the Baseline visit may be enrolled in the study

DETAILED DESCRIPTION:
Phase I/II multicenter, open-label, single-arm trial in patients to evaluate the safety and effect of NECVAX-NEO1 administered in combination with PD-1/PD-L1 mABs in patients with solid tumors. Patients with solid tumors who will be treated with approved standard of care (SoC) PD-1 or PD-L1 monoclonal antibody inhibitor therapy, and who after starting treatment with PD-1/PD-L1 inhibitor reached either Stable Disease (SD) or Partial Response (PR) (Cohort 1) or PD (Cohort 2) according to RECIST 1.1 and iRECIST assessed at the Baseline visit may be enrolled in the study.

Personalised NECVAX-NEO1 is an oral, bacteria-based therapeutic vaccine that incorporates a sequence of patient-specific neoantigens selected by the NEC Immune Profiler. It is designed to stimulate the immune system of patients in order to induce a T-cell response that is able to specifically recognize and destroy tumor cells based on the patient's own neoantigens. NECVAX-NEO1 will be manufactured as a patient-specific Investigational Medicinal Product (IMP) for add-on therapy to the SoC PD-1/PD-L1 inhibitor therapy.

For each patient, the trial will consist of:

* Screening visit: To evaluate patients for inclusion in the trial. The patient signs the informed consent form (ICF), eligibility is confirmed, and a biopsy is taken to start manufacturing of the personalized NECVAX-NEO1.
* Induction period. This is the SoC treatment period, during which treatment with PD-1/PD-L1 inhibitor therapy is started. This is approximately 8 to 12 weeks, depending on the type of PD-1/PD-L1 inhibitor used. The neoantigen selection and manufacturing of the personalized NECVAX-NEO1 takes place during the induction period.
* Baseline visit. At this visit, when the personalized NECVAX-NEO1 treatment is available and the RECIST/iRECIST tumor assessment is performed by magnetic resonance imaging (MRI) or computed tomography (CT) scan, eligibility will be re-confirmed, after which the patient will be assigned to either Cohort 1 (SD or PR according to RECIST 1.1) or Cohort 2 (PD according to RECIST 1.1).
* Treatment period of up to 24 weeks which will mark the addition of new therapy to existing therapy, i.e., prime and booster administrations of NECVAX-NEO1 in addition to PD-1/PD-L1 inhibitor.
* Post-treatment Follow-up period of 4 weeks, with an End of Treatment (EoT) visit at Week 28.
* After the EoT (Week 28), a Long-Term Safety Monitoring Period, following the administration of a genetically modified organism, will occur for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to understand and follow instructions during the trial.
2. Patients able and willing to give written informed consent (signed and dated).
3. Male or female patients.
4. Patients aged at least 18 years old at the time of ICF signature.
5. Patients with solid tumors with measurable disease according to RECIST 1.1, planned to be treated with a PD-1 or PDL1 inhibitor as first- or second-line standard of care therapy according to national/institutional guidelines:
6. Patients with tumor or metastasis accessible for guided needle biopsy or resection.
7. Patients with adequate bone marrow function at Screening, confirmed at Baseline, including:

   1. absolute neutrophil count (ANC) ≥1.5 × 109/L; patients with documented benign cyclical neutropenia are eligible if white blood cell count is ≥1.5 × 109/L, with ANC ≥1.0 × 109/L, leukocytes ≥4.0 × 109/L, and lymphocytes ≥0.6 × 109/L;
   2. platelets ≥ 100 × 109/L;
   3. hemoglobin ≥9 g/dL (may have been transfused);
8. International Normalized Ratio (INR) <1.5 × the upper limit of normal (ULN); patients treated with vitamin K antagonist are eligible if INR <3 (at Screening and confirmed at Baseline).
9. Patients with adequate hepatic function at Screening, confirmed at Baseline, defined by

   1. total bilirubin level ≤1.5 × ULN; patients with documented Gilbert disease are allowed if total bilirubin ≤3 × ULN;
   2. aspartate aminotransferase (AST) level ≤2.5 × ULN, and alanine aminotransferase (ALT) level ≤2.5 × ULN, or, for patients with documented metastatic disease to the liver, AST and ALT levels ≤5 × ULN.
10. Patients with adequate renal function at Screening, confirmed at Baseline, defined by estimated glomerular filtration rate (eGFR) ≥ 30 mL/min using 2021 CKD-EPI creatinine equation (eGFR =142*min(standardized Scr/K, 1)α*max(standardized Scr/K, 1)-1.200 *0.9938Age *1.012 [if female] where K = 0.7 [females] or 0.9 [males], α = -0.241 [females] or -0.302 [males], min = indicates the minimum of Scr/K or 1, and max = indicates the maximum of Scr/K or 1).
11. Patients must be able to undergo MRI or CT scan for tumor follow-up.
12. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
13. Life expectancy of at least 6 months at the time of ICF signature, according to the Investigator's judgement at the time of ICF signature.

Exclusion Criteria:

Medical and surgical history, and diseases

1. History of any disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, based on the Investigator's judgement, provides a reasonable suspicion of a disease or condition that contraindicates the use of the IMP or that might affect the interpretation of the trial results or render the patient at high risk for treatment complications.
2. Symptomatic brain metastasis.
3. Any significant co-morbidity which, according to the Investigator's judgement, makes patient compliance to trial conditions unlikely.
4. Previous malignant disease (other than the tumor disease for this trial) within the last 5 years (except adequately treated non-melanoma skin cancers and carcinoma in situ of skin, bladder, cervix, colon/rectum, breast, or prostate) unless a complete remission without further recurrence was achieved at least 2 years prior to Screening, and the patient is deemed to have been cured with no additional therapy required or anticipated to be required.
5. Prior organ transplantation, including allogeneic stem cell transplantation.
6. Congenital or any other immunodeficiency syndromes, or any active autoimmune disease that might deteriorate when receiving an immunostimulatory agent, except for:

   1. patients with vitiligo, psoriasis, alopecia not requiring immunosuppressive treatment, are eligible.
   2. administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation), which is acceptable.
7. History of uncontrolled intercurrent illness, including but not limited to uncontrolled hypertension (high blood pressure despite of combination therapy with diuretic/CCB/ACE or ARB).
8. Known prior hypersensitivity to the IMP or any component in its formulations or any other drug scheduled or likely to be given during the trial, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥3).
9. Persisting toxicity related to prior therapy (NCI CTCAE v5.0 Grade >1); however, alopecia, sensory neuropathy Grade ≤2, or other Grade ≤2 AEs not constituting a safety risk based on Investigator's judgement are acceptable.
10. Other severe acute or chronic medical conditions (if there is one of the medical conditions at baseline, the patient should not be treated), including

    1. immune colitis
    2. inflammatory bowel disease
    3. history of severe vomiting or diarrhea not having resolved to Grade 1 at Baseline
    4. immune pneumonitis
    5. pulmonary fibrosis
    6. psychiatric conditions including recent (within the last year) or active suicidal ideation or behavior
    7. laboratory abnormalities that may increase the risk associated with trial participation or trial treatment administration or may interfere with the interpretation of trial results and, in the judgement of the Investigator, would make the patient inappropriate for entry into this trial.
11. History of small intestine resection surgery or other major gastrointestinal surgery
12. Active infection requiring systemic therapy with antibiotics (at both Screening and Baseline).
13. Known history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome or multi-drug resistant gram-negative bacteria.
14. Patients with increased anesthesiological risk (e.g. known or predicted difficult airway) if general anesthetic is required.
15. Patients with increased bleeding risk (e.g. coagulopathies) and patients on anticoagulants.
16. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at Screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody Screening test positive).
17. Women who are pregnant or breastfeeding, or women of childbearing potential (defined as any woman who is not surgically sterile with a hysterectomy and/or bilateral oophorectomy or ≥ 12 moths of amenorrhea and at least 50 years of age) not willing to use highly effective methods of birth control up to 6 months after the last dose of IMP. Males of child-bearing potential not willing to use a highly effective method of birth control to avoid pregnancy with any partner during the study and until 90 days after the last dose of IMP
18. Known history of drug/substance abuse. Prior and concomitant medication
19. Live vaccines within 30 days prior to trial treatment.
20. Treatment in any other clinical trial medication within 30 days, before Screening.
21. Any other condition or treatment that, in the opinion of the Investigator, might interfere with the trial.
22. Current drug or substance abuse.
23. Chronic concurrent therapy within 2 weeks before the trial treatment or expected during the trial treatment period with:

    1. corticosteroids (except systemic corticosteroids up to 10 mg prednisolone or equivalent daily dose [oral, intramuscular, or intravenous]).
    2. immunosuppressive agents.
    3. antibiotics.
    4. any other anticancer therapy or concurrent anticancer treatment (except for other checkpoint inhibitors in combination with the anti-PD-1 or anti-PD-L1 monoclonal antibody), for example, cytoreductive therapy, radiotherapy with the exception of palliative short course, limited field (i.e., ≤10 fractions and ≤30% bone marrow involvement or per institutional standard) radiotherapy, which may be administered during the trial. However, IMP dosing must be suspended at least 14 days prior to the start of radiotherapy and must not be resumed until at least 14 days after the last radiotherapy fraction, cytokine therapy, except for erythropoietin.

    Other
24. Inability to understand the Protocol requirements, instructions and trial-related restrictions, the nature, scope, and possible consequences of the trial.
25. Unlikely to comply with the Protocol requirements, instructions, and trial-related restrictions (e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial).
26. Legal incapacity or limited legal capacity.
27. Any condition which results in an undue risk for the patient during the trial participation according to the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Up to week 24 plus 24 months
  AEs listed including system organ class, preferred term, severity, causality and other possibly relevant information. Frequency tables (including both patient and event counts) by System Organ Class (SOC) and preferred term (in number and percentage)
Serious Adverse Events | Up to week 24 plus 24 months
  Serious AEs listed including system organ class, preferred term, severity, causality and other possibly relevant information. Frequency tables (including both patient and event counts) by System Organ Class (SOC) and preferred term (in number and percentage)
Change from Baseline in Laboratory Parameters | Up to week 24 plus 24 months
  Laboratory Parameter Units
Change from Baseline in Electrocardiograms | Up to 24 weeks plus 24 months
  ECG QT interval

SECONDARY OUTCOMES:
Antitumor activity | Up to 24 weeks
  Changes in ctDNA
Objective Response Rate | Up to Week 24 plus 24 months
  Proportion of patients having a best overall response (BOR) of complete response (CR) or partial response (PR) relative to baseline or screening visit
Progression free survival | Up to 24 weeks plus 24 months
  Time from first NECVAX-NEO1 administration to the first of progressive disease (PD) or death
Time to progression | Up to 24 weeks plus 24 months
  Time from first NECVAX-NEO1 administration to PD
Overall survival | Up to 24 weeks plus 24 months
  Time from first NECVAX-NEO1 administration to death

OTHER OUTCOMES:
Tumor immune biomarker | Week 24 compared to Screening
  Number of intratumoral T-cells
Immune response | Up to week 24
  Immune response and pre-existing T-cell pool determined by Enzyme Linked Immuno Spot (ELISpot)
Intestinal microbiome | Up to week 24
  Perentage of bacteria species

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (3):
  - Charité, Berlin
  - NCT, Heidelberg
  - Comprehensive Cancer Center, Munich
- National Cancer Center, Vilnius, Lithuania
- Spain (4):
  - Institut Catala d'Oncologia, Barcelona
  - Vall d'Hebron, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - CHUS Santiago de Compostela, Santiago de Compostela